CLINICAL TRIAL: NCT07135037
Title: Efficacy of L- Arginine Versus Sildenafil in Management of Idiopathic Oligohydramnios
Brief Title: Comparison Between Treatments of Oligohydramnios
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, Ibtesam Teleb Mohamed Yousef Gadalla, principle investigator, Kafrelsheikh University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KFSIRB200-329
Record Dates: First submitted 2025-06-09; First posted 2025-08-21 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2024-09

CONDITIONS: Oligohydramnios
MeSH Terms: conditions — Oligohydramnios | interventions — Sildenafil Citrate; Arginine; Tablets

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- sildn arm (Active Comparator): In this group, participants receive sildenafil 25 mg thrice a day. then amniotic fluid index is measured every week to measure its improvement. After delivery, APGAR will be measured. As well as, whether the fetus entered the NICU or not will be recorded.
  Interventions: Drug: Sildenafil 25 MG
- L- argin arm (Active Comparator): In this group, participants receive L- arginine 1000 mg thrice a day. then amniotic fluid index is measured every week to measure its improvement. After delivery, APGAR will be measured. As well as, whether the fetus entered the NICU or not will be recorded.
  Interventions: Drug: L-Arginine, 1000 Mg Oral Tablet

INTERVENTIONS:
Drug: Sildenafil 25 MG — Sildenafil is a vasodilator drug which improve blood supply to placenta.Therefore, it should improve idiopathic oligohydramnios.
  Other Names: Viagra
  Arms: sildn arm
Drug: L-Arginine, 1000 Mg Oral Tablet — Aminoacid with vasodilator property which improve blood supply to placenta.Therefore, it should improve idiopathic oligohydramnios.
  Other Names: L- arginine
  Arms: L- argin arm

SUMMARY:
Based on previous studies, Both sildenafil and L-arginine helped to improve idiopathic oligohydramnios.

In this study, Level of improvment of oligohydramnios will be compared. As well as, NICU admission to neonates of pregnancies complicated by idiopathic oligohydramnios. The end goal is to help physicians use the best drug for their patients.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women with gestational age between 26-37 weeks
* Pregnant women whose age is < 35 years
* Woman with other indication for elective caesarean section.
* Women carrying a single fetus with no major anomalies.
* Initial amniotic fluid index <8cm determined by reliable pelivabdominal ultrasound.

Exclusion Criteria:

* Women complaining of other obstetric disorder such as, PPROM, preeclampsia, or diabetes.
* Women with chronic illness such as, chronic hypertension, autoimmune disease or kidney disease.
* Women who received other treatments for oligohydramnios in current pregnancy.
* Women who smoke.
* Fetuses with major congenital anomaly.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 40 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-09-15 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Improvement of amniotic fluid index | two hours before cesarean section
  Amniotic fluid index level measured before delivery.

SECONDARY OUTCOMES:
NICU admission | first day after delivery
  NICU admissions rate of the neonates in the study
APGAR score | 5 minutes after delivery
  measuring APGAR score for the neonates in the study

CONTACTS AND LOCATIONS:
Overall Officials: Dalia S Zolfakar, PHD, Study Director — daliasamir94@gmail.com
Locations (2):
- Egypt (2):
  - Kafrelsheikh University Hospital, Kafr ash Shaykh, Kafrelsheikh
  - Kafrelsheokh university hospital, Kafr ash Shaykh, Kafrelsheikh

IPD SHARING:
Plan to Share IPD: Undecided